CLINICAL TRIAL: NCT02322294
Title: A Double-Blind, Placebo-Controlled, Parallel Study to Investigate the Effects of 8 Weeks Use of Glucodia™ on Glucose Parameters, Triglycerides and Body Weight as Compared to Placebo
Brief Title: Investigating the Effects of Glucodia™ on Glucose Parameters, Triglycerides and Body Weight
Acronym: 14GGHF
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: KGK Science Inc. (Industry)
Collaborators: Fuji Oil Co. Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: 14GGHF
Record Dates: First submitted 2014-12-17; First posted 2014-12-23 (Estimated); Last update posted 2016-06-09 (Estimated); Status verified 2016-06

CONDITIONS: Glucose Parameters; Triglycerides; Body Weight
Keywords: Protein; mung bean; glucose; triglycerides; insulin; body weight,; DXA scan
MeSH Terms: conditions — Body Weight; Insulin Resistance

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Glucodia™ (Experimental)
  Interventions: Dietary Supplement: Glucodia™
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Glucodia™
  Arms: Glucodia™
Other: Placebo
  Arms: Placebo

SUMMARY:
This study is investigating the effects of 8 weeks of supplementation with Glucodia™, on glucose parameters, triglycerides and body weight as compared to a placebo. Half of the subjects will be administered Glucodia™, while the other half will receive placebo.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female adults, aged 21 to 45 years
* BMI of 25 kg/m2 to 40 kg/m2 (inclusive)
* Subjects with Fasting Plasma Glucose 5.56mmol/L to 6.94mmol/L (100mg/dL-125mg/dL) AND EITHER Fasting Insulin 60 pmol/L to 180 pmol/L OR Triglycerides 1.36mmol/L to 3.39 mmol/L (120mg/dL-300mg/dL)
* Subject is not of child bearing potential. Defined as females who have had a hysterectomy or oophorectomy, bilateral tubal ligation or are post-menopausal (natural or surgically with > 1 year since last menstruation).

OR Female subject of childbearing potential must agree to use a medically approved method of birth control and have a negative urine pregnancy test result. Acceptable methods of birth control include: Hormonal contraceptives including oral contraceptives, hormone birth control patch (Ortho Evra), vaginal contraceptive ring (NuvaRing), injectable contraceptives (Depo-Provera, Lunelle), or hormone implant (Norplant System), Double-barrier method (condoms with spermicide or diaphragm with spermacide), Non-hormonal intrauterine devices, Vasectomy of partner, Non-heterosexual lifestyle

* Subjects who have no plans to change their smoking habits during the trial period.
* Subjects who are normally active and are deemed to be healthy by the Medical Director
* Subjects who agree to maintain their current level of activity throughout the trial period.
* Subjects who agree to maintain their current dietary habits throughout the trial period.
* Subjects who have given voluntary, written, informed consent to participate in the study.

Exclusion Criteria:

* Subjects who are pregnant, breastfeeding or planning on becoming pregnant throughout the course of the study.
* Subjects with Fasting Glucose < 5.56 mmol/L or > 6.94 mmol/L
* Subjects with Fasting Plasma Glucose 5.56 mmol/L to 6.94 mmol/L who DO NOT have EITHER Fasting Insulin 60 pmol/L to 180 pmol/L OR Triglycerides 1.35 mmol/L to 3.39 mmol/L
* Subjects with BMI < 25 kg/m2 or > 40 kg/m2
* Subjects who have experienced weight loss or gain of greater than 4.5 kg (approximately 10 lbs) in the past 3 months
* Subjects with uncontrolled hypertension ( ≥ 140 mmHg)
* Subjects with any major diseases of the cardiovascular, renal, hepatic, gastrointestinal, pulmonary or endocrine systems
* History of or current diagnosis of any cancer (except for successfully treated basal cell carcinoma) diagnosed less than 5 years prior to screening. Subjects with cancer in full remission more than 5 years after diagnosis are acceptable
* Subjects with neurological disorders or significant psychiatric illnesses
* Subjects with unstable thyroid disease
* Subjects who are immuno-compromised (HIV positive, on anti-rejection medication, rheumatoid arthritis)
* Subjects who have taken any medication or natural health products intended for the management of diabetes, dyslipidemia or body weight within 3 months of randomization.
* Subjects who use illicit drugs or have a history of alcohol or drug abuse within the past 6 months
* Subjects who currently consume greater than 2 standard alcoholic drinks per day.
* Subjects who have participated in a clinical research trial within 30 days prior to randomization.
* Subjects with an allergy or sensitivity to the investigational product ingredient.
* Subjects who are cognitively impaired and/or who are unable to give informed consent
* Subjects who have abnormal laboratory results or any other medical or psychological condition which, in the opinion of the Principle Investigator, may adversely affect the subjects ability to complete the study or its measures or which may pose significant risk to the subject

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2015-01; Primary Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Change in glucose response to 2-hour oral glucose tolerance test (OGTT) in subjects taking Glucodia™ versus Placebo | Baseline and week 8
  Assessed by the change in the area under the curve in glucose response

SECONDARY OUTCOMES:
Change in insulin response to 2-hour oral glucose tolerance test (OGTT) in subjects taking Glucodia™ versus Placebo | Baseline and week 8
  Assessed by the change in the area under the curve in insulin response
Change in fasting glucose in subjects taking Glucodia™ versus Placebo | Baseline, week 4 and week 8
Change in fasting insulin in subjects taking Glucodia™ versus Placebo | Baseline, week 4 and week 8
Change in HOMA-IR in subjects taking Glucodia™ versus Placebo | Baseline, week 4 and week 8
Change in adiponectin levels in subjects taking Glucodia™ versus Placebo | Baseline, week 4 and week 8
Change in lipid panel levels in subjects taking Glucodia™ versus Placebo | Baseline, week 4 and week 8
  Lipid panel includes total cholesterol, triglycerides, HDL, LDL, free fatty acids and non-esterified fatty acids
Change in body composition in subjects taking Glucodia™ versus Placebo | Baseline, week 4 and week 8
  Assessed via DXA scan
Change in body composition in subjects taking Glucodia™ versus Placebo | Baseline, week 4 and week 8
  Assessed via circumference measurements of the arm, thigh, hip and waist and the hip to waist ratio
Change in body weight in subjects taking Glucodia™ versus Placebo | Baseline, week 4 and week 8
Change in appetite in subjects taking Glucodia™ versus Placebo | Baseline, week 4 and week 8
  Assessed using a Satiety VAS scale questionnaire

OTHER OUTCOMES:
Changes in Vital Signs in subjects taking Glucodia™ versus Placebo | Screening, Baseline, week 4, week 8
  Blood Pressure and Heart Rate
Changes in Blood Hematology and Clinical Chemistry in subjects taking Glucodia™ versus Placebo | Screening, Baseline, week 4 and week 8
  CBC, electrolytes, creatinine, AST, ALT, GGT, bilirubin, HbA1c, BUN, total protein, albumin, globulin and calcium

CONTACTS AND LOCATIONS:
Overall Officials: Tetyana Pelipyagina, MD, Principal Investigator — KGK Science Inc.
Locations (1):
- KGK Synergize Inc., London, Ontario, Canada